CLINICAL TRIAL: NCT05419986
Title: Are Epigenetic Biomarkers an Indicator of the Severity of Addiction in Active Opiate Abusers? A Pilot Study
Brief Title: Epigenetic Biomarker for Opioid Use Disorder
Acronym: EBIOMOUD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: stop due to lack of funds
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 8484
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Opioid Use Disorder; Addiction
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-opioid users (Other)
  Interventions: Genetic: Blood collection
- Active opioid users (Other)
  Interventions: Genetic: Blood collection

INTERVENTIONS:
Genetic: Blood collection — Molecular monitoring by measure of DNA methylation levels in blood samples collected by fingerstick blood drops, as opposed to veinous phlebotomy

SUMMARY:
Study rationale Opioid use disorder (OUD) is a chronic and severe condition, defined by problematic opioid use, which results from interactions among sociological factors, psychiatric symptoms and life experiences, altogether determining OUD severity.

Recently, behavioral epigenetics has emerged as a possible strategy to help identify molecular mechanisms that may explain how these various interactions result in dysregulations affecting gene expression, brain function, and, ultimately, emotional regulation.

Here the investigators propose a pilot study as a first step towards a larger multidisciplinary project whose goal will be to characterize simultaneously major psychiatric and social factors in individuals with OUD, across a wide range of disease severity. In the present pilot study, the investigators propose to first characterize technical feasibility of the molecular investigations proposed in these 2 projects.

OUD severity The severity of OUD is well defined in the DSM-5 (2013), with 3 categories, from mild to severe, on the basis of the number of dimensional criteria met by patients (among 11 criteria). These criteria relate to the following main aspects: tolerance, the need to increase the amount of drugs to avoid withdrawal; psychic and physic withdrawal in case of substance discontinuation; social and interpersonal consequences of drug use; biological and psychic consequences of use; and craving, the irrepressible need to consume1. Here, the investigators postulate that molecular adaptations detected in the blood of OUD patients may represent biomarkers of this severity.

Epigenetic blood biomarkers A main limitation for conducting peripheral blood biomarker investigations in active opioid abusers comes from the fact that phlebotomies are reputedly difficult & potentially iatrogenic in these subjects, as they associate with external cues and trigger internal states that are closely related to drug consumption. To overcome this difficulty, we propose to test the hypothesis that sufficient DNA amounts can be recovered from fingerstick blood drops (corresponding to capillary blood, similar to sugar testing) to generate robust and reliable DNA methylation measures in the full human epigenome. In other words, the investigators assume that DNA methylation can be measured using capillary blood.

Objectives The investigators will first investigate in healthy volunteers whether the method consisting in collecting and analyzing small DNA amounts from capillary blood (fingerstick blood drops) retrieves DNA methylation measures for a number of CG dinucleotide sites (where DNA methylation occurs in the mammalian genome) that is comparable to that classically observed using veinous blood (phlebotomy). Second, the investigators will test the feasibility of measuring DNA methylation using capillary blood samples collected from patients with OUD.

To this purpose, the investigators propose to collect veinous and capillary blood samples from healthy volunteers, and capillary blood from opioid users.

ELIGIBILITY:
Inclusion criteria

First step:

* Healthy volunteers subjects (men or women) at least 18 years old
* Subjects affiliated to a social health insurance scheme
* Able to understand the objectives and risks of the research and to give dated and signed informed consent
* Without any drug use except tobacco consumption and/or occasional alcohol consumption (defined by not more than 21 drinks per week for men and note more than 14 drinks per week for women)

Second step :

* Subjects (Male or female) active opioid users at least 18 years old
* Subjects affiliated to a social health insurance scheme
* Able to understand the objectives and risks of the research and to give dated and signed informed consent

Exclusion criteria:

Impossibility of giving information to the subject (subject in an emergency situation, difficulties in understanding the subject, etc.)

* Subjects in an exclusion period (determined by a previous or current study),
* Subjects already participating to another study with an investigational product
* Subjects under court protection (patients deprived of freedom because of a judicial measure)
* Subjects under guardianship or curatorship
* Subjects with severe psychiatric disease (bipolar disorder, schizophrenia, chronic psychotic disorder) Authorized and/or prohibited drugs/treatments
* No treatment or drug use will be authorized for healthy volunteers during the first step study (with exceptions for occasional alcohol or tobacco use).
* All treatments will be authorized for the step 2 study in opioid users.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Comparison of DNA methylation between fingerstick drop samples and venous samples | 1 day
  Quantitative description of the number of CG dinucleotide sites where sufficient coverage can be obtained (>5X) in blood samples collected by fingerstick blood drops versus venous blood samples, using Reduced Representation Enzymatic Methylation Sequencing (RREMseq), in healthy volunteers and in subjects with OUD.

SECONDARY OUTCOMES:
Correlation between Opioid Use Disorder (OUD) severity and DNA methylation in capillary blood samples of patients with OUD | 1 day
  1. Quantitative description of the number of subjects with severe OUD (meeting at least 6 out of 11 DSM-5 criteria) / without severe OUD (less than 6 criteria)
  2. Preliminary quantitative description of DNA methylation levels in capillary blood samples from patients with / without severe OUD

CONTACTS AND LOCATIONS:
Overall Officials: Laurence LALANNE, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Laurence LALANNE, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided